CLINICAL TRIAL: NCT00694473
Title: Continuous Glucose Monitoring With a Subcutaneous Sensor During Critical Illness and Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Abbott Diabetes Care (Industry)
Responsible Party: Principal Investigator, Steven J. Russell, MD, PhD, Assistant in Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007P-002178
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Results first posted 2017-10-06 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-02

CONDITIONS: Critical Illness
Keywords: hyperglycemia; hypoglycemia; insulin; critical illness; intensive insulin therapy; continuous glucose monitoring; CGM; interstitial fluid glucose; intensive care unit; Blood glucose
MeSH Terms: conditions — Critical Illness; Hyperglycemia; Hypoglycemia; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Freestyle Navigator (Experimental): Continuous monitoring with the Freestyle Navigator for 72 hours or until discharge from the ICU
  Interventions: Device: Freestyle Navigator

INTERVENTIONS:
Device: Freestyle Navigator — Continuous glucose monitoring with the Freestyle Navigator for 72 hours or until discharge from the ICU

SUMMARY:
We hypothesize that measurements of interstitial fluid (ISF) glucose by the FreeStyle Navigator (Abbot Diabetes Care), a continuous glucose monitoring system, will correlate with blood glucose (BG) values in surgical and ICU patients with a clinically useful degree of accuracy.

DETAILED DESCRIPTION:
Critically ill patients treated with intensive insulin therapy will be monitored for up to 72 hours with the Freestyle Navigator continuous glucose monitor. The device display will be disabled so that continuous glucose monitoring results will not be available to care givers, although low (<60 mg/dL) and high (>250 mg/dL) threshold audio alarms will be enabled. Blood glucose monitoring will be performed according to the usual practice for patients treated with intensive insulin therapy in each intensive care unit, except that additional blood glucose measurements will be performed in response to Freestyle Navigator threshold alarm. All blood glucose management decisions will be made according to intensive insulin therapy protocol in each unit. Freestyle Navigator data will be downloaded from the device after each subject has completed the monitoring period. Blood glucose values obtained in the course of usual care, or in response to Freestyle Navigator threshold alarms, will be compared with time-matched Freestyle Navigator values to assess device accuracy and alarm sensitivity and specificity.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the general surgical ICU (SICU), medical ICU (MICU), cardiac surgery intensive care unit (CSICU), or neurological intensive care unit (NeuroICU), are being treated with IIT, and have an arterial line in place
* Patients scheduled for open cardiac surgery or craniotomy that have diabetes mellitus or will be given high dose glucocorticoids. All of these patient will have an arterial line placed at the time of surgery as a part of their usual care

Exclusion Criteria:

* Age less than 18 years
* Enrollment in another clinical trial that modifies their glucose management (e.g. trial of modified IIT algorithm or modified glucose monitoring regimen)

In order to obtain adequate representation of patients with physiological alterations that might decrease correspondence between blood and ISF glucose, we will recruit 50 subjects in each of five groups:

1. Patients undergoing craniotomy who are either diabetic or will be given high dose corticosteroids
2. Diabetic patients undergoing open cardiac surgery
3. Patients admitted to one of the participating ICUs with an arterial line in place and receiving IIT who are vasopressor dependent, defined by continuous infusion of at least 60 mg/min phenylephrine, 5 mg/min norepinephrine, or 10 mg/kg/min of dopamine, or any combination of two agents for at least 90 continuous minutes in the last 8 hours
4. Patients admitted to one of the participating ICUs with an arterial line in place and receiving IIT with pitting peripheral or dependent edema, defined by the persistence of pitting to at least 5 mm depth for 5 seconds after pressure is applied to a dependent area of the trunk or two limbs.
5. Critically ill patients admitted to one of the participating ICUs with an arterial line in place and receiving IIT who do not fall into groups 1-4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2008-06; Primary Completion 2010-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J. Russell, M.D., Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Freestyle Navigator
Started | 76 (Aug 2008)
Completed | 69 (Dec 2010)
Not Completed | 7

BASELINE CHARACTERISTICS:
Population: 76 were enrolled, analysis was completed for 69
Arm/Group | Freestyle Navigator
Number analyzed (Participants) | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 38
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 69

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity of Navigator Threshold Alarms for Hypoglycemia (<60 mg/dl).
Time Frame: 72 hours
Population: This measure was not calculated as we did not have sufficient data to calculate sensitivity (not enough hypoglycemia) and discordant BG check times to calculate specificity.
Arm/Group | Freestyle Navigator
Number analyzed (Participants) | 0

2. Secondary Outcome: Sensitivity and Specificity of Navigator Threshold Alarms for Hyperglycemia (>240 mg/dl).
Time Frame: 72 hours
Population: This measure was not calculated as we did not have sufficient data to calculate sensitivity and inappropriate BG check times to calculate specificity and few trends towards hyperglycemia
Arm/Group | Freestyle Navigator
Number analyzed (Participants) | 0

3. Secondary Outcome: Accuracy of Navigator CGM as Compared to Reference Blood Glucose Values
Description: Mean Absolute Relative Difference (MARD) of Navigator CGM compared with reference blood glucose values
Time Frame: 72 hours
Measure: Mean (Full Range); unit: percent absolute relative difference
Arm/Group | Freestyle Navigator
Number analyzed (Participants) | 69
percent absolute relative difference | 14.5 [13.0 to 16.0]

4. Secondary Outcome: Sensitivity and Specificity of Navigator Projected Low Blood Sugar Alarm Criteria Calculated for Events Defined by a Low Reference BG Value (< 60 mg/dL)
Time Frame: 72 hours
Population: as for outcome 1
Arm/Group | Freestyle Navigator
Number analyzed (Participants) | 0

5. Secondary Outcome: Sensitivity and Specificity of Navigator Projected High Blood Sugar Alarm Criteria Calculated for Events Defined by a High Reference BG Value (> 250 mg/dl)
Time Frame: 72 hours
Population: as for outcome 2
Arm/Group | Freestyle Navigator
Number analyzed (Participants) | 0

6. Secondary Outcome: Percentage of Readings in Different Blood Sugar Ranges as Shown by Point of Care Testing:
Description: Percentage of readings in different blood sugar ranges as shown by point of care testing:
  < 60 mg/dl 61-120 mg/dl 121-180 mg/dl 181-240 lmg/dl >240 mg/dl
Time Frame: 72 hours
Measure: Number; unit: percentage of readings
Arm/Group | Freestyle Navigator
Number analyzed (Participants) | 69
percentage of readings
  <60mg/dl | 10
  61-120mg/dl | 23
  121-180mg/dl | 41
  181-240mg/dl | 12
  >240mg/dl | 14

7. Secondary Outcome: Navigator CGM Accuracy by Category
Description: Mean Absolute Relative Difference (MARD) between the Navigator CGM and reference blood glucose values by category (1, Neurosurgery; 2, Cardiac Surgery; 3, Hypotensive/Vasopressor; 4, Edema; 5, None of the Above)
Time Frame: 72 hours
Population: MARD by category (1, Neurosurgery; 2, Cardiac Surgery; 3, Hypotensive/Vasopressor; 4, Edema; 5, None of the Above)
Measure: Mean (Standard Deviation); unit: percent absolute relative difference
Arm/Group | Freestyle Navigator
Number analyzed (Participants) | 69
percent absolute relative difference
  Neurosurgery | 15.1 (12.7)
  Cardiac surgery | 14.3 (14.6)
  Hypotensive/vasopressor | 18.8 (18.6)
  Edema | 9.7 (4.1)
  None | 10.1 (10.0)

ADVERSE EVENTS:
Time Frame: 72 hours
Arm/Group | Freestyle Navigator
All-Cause Mortality (participants affected / at risk) | 1/69
Serious Adverse Events (participants affected / at risk) | 0/69
Other Adverse Events (participants affected / at risk) | 5/69
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Freestyle Navigator (N=69)
Bleeding at Insertion Site (Injury, poisoning and procedural complications) | 4 (4) — Bleeding at the insertion site of the subcutaneous sensor
Culture proven bacteremia (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Analysis used recalibrated data from Abbot; possible bias. Time of A-line removal was not always documented; estimate of arterial vs. venous POC reference BGs is estimated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No